CLINICAL TRIAL: NCT01364311
Title: Treatment of Dry Eye With Supplements
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhofer, MD, Ass.-Prof., Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-120111
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2014-11

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes; Dietary Supplements; Vitamac® Tag and Nacht capsules; Lutein; Vitamin C; Zinc; ginkgo biloba; Flavinoids; Fishoil; Zeaxanthin; Vitamin E; Copper; Selen; Alpha Lipon acid; Break up time (BUT); Improvement of subjective symptoms of dry eye syndrome; Visual Acuity; Tear film osmolarity; OSI (Objective Scattering Index); Schirmer I test; Staining of the cornea with fluorescein; Impression cytology; Tear cytokines/chemokines; Data from patient diary how often Hylo-Comod® eye drops were used
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Vitamac® Tag and Nacht capsules — Vitamac® Tag und Nacht Kapseln: Dosage 1 capsule Vitamac® Tag per day ingested in the morning, 1 capsule Vitamac® Nacht per day ingested in the evening.
  Vitamac® Tag: Lutein 12mg, Vitamin C 300mg, Zinc 10mg, ginkgo biloba 10mg, Flavinoids 25mg, Fishoil 300mg, administered for 12 weeks Vitamac® Nacht: Zeaxanthin 5mg, Vitamin E 60mg, Copper 1mg, Selen 20µg, Ginkgo Biloba 10mg, Flavinoids 25mg, Alpha Lipon acid 150mg), administered for 12 weeks

SUMMARY:
Dry eye syndrome (DES) is a highly prevalent ocular condition inducing an inflammatory response on the ocular surface. Common symptoms include ocular discomfort, visual impairment and instability of the tear film with potential damage to the ocular surface.

In addition, an intact tear film is important to provide a smooth optical surface, to act as a barrier to pathogens, to nourish the epithelial cells of the ocular surface and to prevent exsiccation. Alterations in the tear film composition, which can have their origin in several conditions, lead to tear film hyperosmolarity or instability resulting in DES.

Regardless of the cause of DES, chronic dryness of the ocular surface leads to an increased susceptibility to oxidative stress, which is triggered by reactive oxygen species (ROS). This results in cell damage and activation of the immune system, keeping up inflammatory processes . In order to prevent ROS damage, several micronutrients such as vitamin C, E, and certain carotenoids, omega-3 free fatty acids, flavonoids and minerals have been used because of their antioxidant capacities.

Based on this knowledge the potential of these antioxidant dietary supplements has been discussed as a treatment option for DES. Preliminary data support the hypothesis that antioxidant supplementations, in particular, supplementation with omega 3 fatty acids may be beneficial for patients with DES.

The purpose of the present study is to test the hypothesis that treatment with dietary supplements improves subjective and objective symptoms of DES.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* History of dry eye syndrome for at least 3 months
* Tear Break Up Time (BUT) < 10 seconds or Schirmer I test < 7 mm
* At least 2 symptoms of dry eye syndrome (foreign body sensation, burning, photophobia, blurred vision, pain, itching)
* -Normal ophthalmic findings except dry eye syndrome

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Wearing of contact lenses
* Intake of dietary supplements in the 3 months preceding the study
* Glaucoma
* Treatment with corticosteroids in the 4 weeks preceding the study
* Topical treatment with any ophthalmic drug except topical lubricants in the 4 weeks preceding the study
* Ocular infection or inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Improvement of subjective symptoms of dry eye syndrome | 12 weeks
Break up time (BUT) | 12 weeks

SECONDARY OUTCOMES:
Visual Acuity | 12 weeks
Tear film osmolarity | 12 weeks
OSI (Objective Scattering Index) | 12 weeks
Schirmer I test | 12 weeks
Staining of the cornea with fluorescein | 12 weeks
Impression cytology | 12 weeks
Tear cytokines/chemokines | 12 weeks
Data from patient diary how often Hylo-Comod® eye drops were used | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Schmidl, MD, Principal Investigator — Department of Clinical Pharmacology,Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Austria